CLINICAL TRIAL: NCT01081184
Title: Neurotrophins Implications in Primary Sjögren Syndrome
Acronym: Neuro-SGSp
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I08010
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2010-03

CONDITIONS: Primary Sjögren Syndrome
Keywords: primary Sjögren syndrome; neurotrophins; B cell; sicca syndrome; T cell
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- primary Sjögren syndrome
  Interventions: Biological: blood sample
- Healthy volunteers
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sample for determination of seric and lymphocytic NT profile will be added to a standard biological analysis done for pSS follow- up
  Other Names: Salivary sicca syndrome will be evaluated.; Saliva fluid will be collected.; Ocular sicca syndrome will be evaluated.; A conjonctival cytological impression will be done.

SUMMARY:
Neurotrophins (NTs) constitute a family of growth factors, which regulated differentiation, proliferation, and survival of both neuronal cells and astrocytes. In recent years, several studies have provided evidences that the cellular effects of NGF " Nerve Growth Factor ", BDNF " Brain-Derived Neurotrophic Factor " and NT-3 are not limited to the nervous system. Indeed, neurotrophins and their receptors are widely expressed on non neuronal cells. Data concerning the implication of NTs and their receptors in the immune system maturation and in the regulation of normal and pathological immune responses are numerous and suggest the existence of a specific "neuro-immunomodulation" through these neuropeptides.

The aim of the study is to compare Sjögren's syndrome systemic activity to seric, lymphocytic and conjunctival levels of NTs (i.e NGF, BDNF and NT-3). A preliminary study has previously pointed out the link between high BDNF seric levels and Sjögren's systemic activity. The increased levels of BDNF were correlated to T cell activation. A similar correlation between high NGF level and hypergammaglobulinemia was also pointed out.

DETAILED DESCRIPTION:
2 supplementary blood sample for determination of seric and lymphocytic NT profile will be added to a standard biological analysis done for pSS follow- up.

Salivary sicca syndrome will be evaluated with un-stimulated salivary flow rate. Saliva fluid will be collected from NTs levels determination (ELISA). Ocular sicca syndrome will be evaluated by Schirmer tests and Lissaline green test. A conjunctival cytological impression will be done in order to determine NTs conjunctival production by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

Arm : primary Sjögren syndrome:

* All patients must fulfill the revised criteria for primary Sjögren syndrome.
* Age of entry into the study ≥ 18 yrs.
* Affiliated or profit patient of a social security system.
* Informed consent signed up.

Arm : healthy volunteers:

* All patient free of autoimmune disease.
* Age of entry into the study ≥ 18 yrs.
* Affiliated or profit patient of a social security system.
* Informed consent signed up.

Exclusion Criteria:

* Patient with psychiatric disorders not related with antiphospholipid syndrome and / or cerebral complication of SGSp.
* Addictive behaviors (alcoholism, cocaine or opioid abuse).
* Patient with anti-depressive drugs.
* Patient with concurrent malignancy
* Pregnancy
* Patients under measure of maintenance of justice.
* Patients unable to understand or to participate to the study.
* Child and major patients making the object of a measure of lawful protection.
* Patients deprived of freedom.

Exclusion criteria for control group

* Autoimmune disease.
* Steroid treatment (>20 mg/day).
* Immunosuppressive treatment.
* Concurrent malignancy.
* Concurrent psychiatric disorders.
* Anti-depressive drugs.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with primary Sjögren syndrome
  People free of disease : healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Lymphocytic levels of NTs (i.e. NGF, BDNF and NT-3) | 1 day
  2 supplementary blood sample for determination of seric and lymphocytic NT profile will be added to a standard biological analysis done for pSS follow- up.

SECONDARY OUTCOMES:
Disease activity score used: ESSDAI; NGF, BDNF and NT3 levels in sera; pSS immunological profile; intensity of sicca syndrome; salivary levels of NTs; conjunctival expression of NTs. | 1 day
  Salivary sicca syndrome will be evaluated with un-stimulated salivary flow rate. Saliva fluid will be collected from NTs levels determination (ELISA). Ocular sicca syndrome will be evaluated by Schirmer tests and Lissaline green test. A conjunctival cytological impression will be done in order to determine NTs conjonctival production by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure FAUCHAIS, MD, Principal Investigator — Limoges UH
Locations (2):
- France (2):
  - Médecine Interne, Limoges
  - Opthalmologie, Limoges